CLINICAL TRIAL: NCT02812680
Title: The Utility of Circulating Tumour Cells and Plasma microRNA Detection to Predict the Response to Treatment in Patients With Esophageal Adenocarcinoma
Brief Title: The Utility of Circulating Tumour Cells and Plasma microRNA in Esophageal Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 15-9303-CE
Record Dates: First submitted 2016-06-14; First posted 2016-06-24 (Estimated); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Esophageal Cancer Patients - Blood Draw: Look at blood samples to assess the use of circulating microRNA (miRNA) and circulating tumour cells (CTC) as biomarkers of cancer and predictive markers for neoadjuvant therapy in patients with Esophageal Adenocarcinoma.
  Interventions: Other: Blood Draw
- Healthy volunteers - Blood Draw: Comparators for the esophageal cancer group
  Interventions: Other: Blood Draw

INTERVENTIONS:
Other: Blood Draw — Blood draw to assess the use of circulating microRNA (miRNA) and circulating tumour cells (CTC) as biomarkers of cancer and predictive markers for neoadjuvant therapy.

SUMMARY:
Circulating microRNA (circ miRNA) and circulating tumor cell (CTC) levels are hypothesized to be associated with response to chemoradiation in patients undergoing treatment for locally advanced esophageal adenocarcinoma.

The goal of this project is to assess the use of circulating microRNA (miRNA) and circulating tumour cells (CTC) as biomarkers of cancer and predictive markers for neoadjuvant therapy.

DETAILED DESCRIPTION:
Recently, different groups have discovered that miRNAs can be detected in body fluids such as plasma, serum or saliva. These cell-free miRNAs are secreted by cells under different forms. Levels of these circulating miRNAs (circ miRNA), like tissue miRNA, were closely related to pathologies and could be used as diagnostic or prognostic tools for several pathologies, including cancer. Furthermore, a recent report showed that circ miRNAs released by tumor cells have the ability to transfer their metastatic potential to nonmetastatic cells. The detection and analysis of circulating miRNA represent a new step towards non-invasive diagnostic screening and early cancer detection.

Circulating tumor cells also hold promise as biological markers, which can be assessed noninvasively. As more than 90% of cancer deaths are associated with metastasis, it is crucial to understand the mechanisms of dissemination of cancer cells. During the past decade, a multitude of techniques have been developed to track down and to characterize CTC. Clinical studies in various cancers reveal the potential of CTC as prognostic and predictive markers. The characterization of CTC will help to design personalized treatment to eradicate the sub-clones of the primary tumour, which give rise to metastasis. Also, the numbers of CTC in patient blood can be followed to monitor the efficacy of the neoadjuvant treatment.

Most of the research in esophageal cancer has been done on squamous cell cancer as this is the dominant cell type worldwide. However, beginning the in 1980s Esophageal Adenocarcinoma (EAC) has increased in frequency such that it now represents 80% of esophageal cancer in North America and Europe. There is an urgent need to develop new techniques and diagnostic tests to combat EAC. By combining circ miRNA and CTC, we not only combine 2 promising clinical biomarkers, we will also be able to access new data that will complement tissue biopsy data. Furthermore, by acquiring a blood sample during various time points of patient treatment, we will be able to create a dynamic CTC and circ miRNA profile.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age
* Patients with Esophageal Adenocarcinoma who will undergo neo-adjuvant therapy with surgical resection.
* Patients with esophageal adenocarcinoma who will be treated with chemotherapy, chemotherapy and radiation or radiation alone OR
* Healthy volunteers who are at least 18 years of age

Exclusion Criteria:

* Patients who are treated with surgery alone for esophageal cancer
* Patients who have a history of invasive cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Esophageal Cancer Patients vs Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Circulating microRNA (miRNA) as biomarkers of cancer and predictive markers for neoadjuvant therapy by using Human miRNA cards | 2 years
Circulating tumour cells (CTC) as biomarkers of cancer and predictive markers for neoadjuvant therapy by using CTC chips | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gail E Darling, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Blot WJ. Esophageal cancer trends and risk factors. Semin Oncol. 1994 Aug;21(4):403-10. PMID 8042037
- [Background] Parkin DM, Bray F, Ferlay J, Pisani P. Global cancer statistics, 2002. CA Cancer J Clin. 2005 Mar-Apr;55(2):74-108. doi: 10.3322/canjclin.55.2.74. PMID 15761078
- [Background] Demeester SR. Epidemiology and biology of esophageal cancer. Gastrointest Cancer Res. 2009 Mar;3(2 Suppl):S2-5. PMID 19461918
- [Background] Davies AR, Gossage JA, Zylstra J, Mattsson F, Lagergren J, Maisey N, Smyth EC, Cunningham D, Allum WH, Mason RC. Tumor stage after neoadjuvant chemotherapy determines survival after surgery for adenocarcinoma of the esophagus and esophagogastric junction. J Clin Oncol. 2014 Sep 20;32(27):2983-90. doi: 10.1200/JCO.2014.55.9070. PMID 25071104
- [Background] Bartel DP. MicroRNAs: genomics, biogenesis, mechanism, and function. Cell. 2004 Jan 23;116(2):281-97. doi: 10.1016/s0092-8674(04)00045-5. PMID 14744438
- [Background] Bartel DP. MicroRNAs: target recognition and regulatory functions. Cell. 2009 Jan 23;136(2):215-33. doi: 10.1016/j.cell.2009.01.002. PMID 19167326
- [Background] Flynt AS, Lai EC. Biological principles of microRNA-mediated regulation: shared themes amid diversity. Nat Rev Genet. 2008 Nov;9(11):831-42. doi: 10.1038/nrg2455. PMID 18852696
- [Background] Esquela-Kerscher A, Slack FJ. Oncomirs - microRNAs with a role in cancer. Nat Rev Cancer. 2006 Apr;6(4):259-69. doi: 10.1038/nrc1840. PMID 16557279
- [Background] Calin GA, Croce CM. MicroRNA signatures in human cancers. Nat Rev Cancer. 2006 Nov;6(11):857-66. doi: 10.1038/nrc1997. PMID 17060945
- [Background] Lawrie CH, Cooper CD, Ballabio E, Chi J, Tramonti D, Hatton CS. Aberrant expression of microRNA biosynthetic pathway components is a common feature of haematological malignancy. Br J Haematol. 2009 May;145(4):545-8. doi: 10.1111/j.1365-2141.2009.07642.x. Epub 2008 Mar 2. No abstract available. PMID 19298586
- [Background] Mitchell PS, Parkin RK, Kroh EM, Fritz BR, Wyman SK, Pogosova-Agadjanyan EL, Peterson A, Noteboom J, O'Briant KC, Allen A, Lin DW, Urban N, Drescher CW, Knudsen BS, Stirewalt DL, Gentleman R, Vessella RL, Nelson PS, Martin DB, Tewari M. Circulating microRNAs as stable blood-based markers for cancer detection. Proc Natl Acad Sci U S A. 2008 Jul 29;105(30):10513-8. doi: 10.1073/pnas.0804549105. Epub 2008 Jul 28. PMID 18663219
- [Background] Park NJ, Zhou H, Elashoff D, Henson BS, Kastratovic DA, Abemayor E, Wong DT. Salivary microRNA: discovery, characterization, and clinical utility for oral cancer detection. Clin Cancer Res. 2009 Sep 1;15(17):5473-7. doi: 10.1158/1078-0432.CCR-09-0736. Epub 2009 Aug 25. PMID 19706812
- [Background] Turchinovich A, Weiz L, Burwinkel B. Extracellular miRNAs: the mystery of their origin and function. Trends Biochem Sci. 2012 Nov;37(11):460-5. doi: 10.1016/j.tibs.2012.08.003. Epub 2012 Sep 1. PMID 22944280
- [Background] Cortez MA, Bueso-Ramos C, Ferdin J, Lopez-Berestein G, Sood AK, Calin GA. MicroRNAs in body fluids--the mix of hormones and biomarkers. Nat Rev Clin Oncol. 2011 Jun 7;8(8):467-77. doi: 10.1038/nrclinonc.2011.76. PMID 21647195
- [Background] Le MT, Hamar P, Guo C, Basar E, Perdigao-Henriques R, Balaj L, Lieberman J. miR-200-containing extracellular vesicles promote breast cancer cell metastasis. J Clin Invest. 2014 Dec;124(12):5109-28. doi: 10.1172/JCI75695. Epub 2014 Nov 17. PMID 25401471
- [Background] Hanahan D, Weinberg RA. Hallmarks of cancer: the next generation. Cell. 2011 Mar 4;144(5):646-74. doi: 10.1016/j.cell.2011.02.013. PMID 21376230
- [Background] Krebs MG, Metcalf RL, Carter L, Brady G, Blackhall FH, Dive C. Molecular analysis of circulating tumour cells-biology and biomarkers. Nat Rev Clin Oncol. 2014 Mar;11(3):129-44. doi: 10.1038/nrclinonc.2013.253. Epub 2014 Jan 21. PMID 24445517
- [Background] Joosse SA, Gorges TM, Pantel K. Biology, detection, and clinical implications of circulating tumor cells. EMBO Mol Med. 2015 Jan;7(1):1-11. doi: 10.15252/emmm.201303698. PMID 25398926
- [Background] Knox JJ, Wong R, Visbal AL, Horgan AM, Guindi M, Hornby J, Xu W, Ringash J, Keshavjee S, Chen E, Haider M, Darling G. Phase 2 trial of preoperative irinotecan plus cisplatin and conformal radiotherapy, followed by surgery for esophageal cancer. Cancer. 2010 Sep 1;116(17):4023-32. doi: 10.1002/cncr.25349. PMID 20533506
- [Background] Underwood TJ, Derouet MF, White MJ, Noble F, Moutasim KA, Smith E, Drew PA, Thomas GJ, Primrose JN, Blaydes JP. A comparison of primary oesophageal squamous epithelial cells with HET-1A in organotypic culture. Biol Cell. 2010 Dec;102(12):635-44. doi: 10.1042/BC20100071. PMID 20843300
- [Background] Ko MA, Zehong G, Virtanen C, Guindi M, Waddell TK, Keshavjee S, Darling GE. MicroRNA expression profiling of esophageal cancer before and after induction chemoradiotherapy. Ann Thorac Surg. 2012 Oct;94(4):1094-102; discussion 1102-3. doi: 10.1016/j.athoracsur.2012.04.145. Epub 2012 Aug 29. PMID 22939244
- [Background] Derouet MF, Liu G, Darling GE. MiR-145 expression accelerates esophageal adenocarcinoma progression by enhancing cell invasion and anoikis resistance. PLoS One. 2014 Dec 31;9(12):e115589. doi: 10.1371/journal.pone.0115589. eCollection 2014. PMID 25551563
- [Background] Underwood TJ, Hayden AL, Derouet M, Garcia E, Noble F, White MJ, Thirdborough S, Mead A, Clemons N, Mellone M, Uzoho C, Primrose JN, Blaydes JP, Thomas GJ. Cancer-associated fibroblasts predict poor outcome and promote periostin-dependent invasion in oesophageal adenocarcinoma. J Pathol. 2015 Feb;235(3):466-77. doi: 10.1002/path.4467. PMID 25345775
- [Background] Mohamadi RM, Besant JD, Mepham A, Green B, Mahmoudian L, Gibbs T, Ivanov I, Malvea A, Stojcic J, Allan AL, Lowes LE, Sargent EH, Nam RK, Kelley SO. Nanoparticle-mediated binning and profiling of heterogeneous circulating tumor cell subpopulations. Angew Chem Int Ed Engl. 2015 Jan 2;54(1):139-43. doi: 10.1002/anie.201409376. Epub 2014 Nov 5. PMID 25377874
- [Background] Tsujiura M, Ichikawa D, Komatsu S, Shiozaki A, Takeshita H, Kosuga T, Konishi H, Morimura R, Deguchi K, Fujiwara H, Okamoto K, Otsuji E. Circulating microRNAs in plasma of patients with gastric cancers. Br J Cancer. 2010 Mar 30;102(7):1174-9. doi: 10.1038/sj.bjc.6605608. Epub 2010 Mar 16. PMID 20234369
- [Background] Resnick KE, Alder H, Hagan JP, Richardson DL, Croce CM, Cohn DE. The detection of differentially expressed microRNAs from the serum of ovarian cancer patients using a novel real-time PCR platform. Gynecol Oncol. 2009 Jan;112(1):55-9. doi: 10.1016/j.ygyno.2008.08.036. Epub 2008 Oct 26. PMID 18954897
- See also: Canadian Cancer Statistics 2010 — http://www.cancer.ca